CLINICAL TRIAL: NCT05041803
Title: A Multicenter, Open-Label, Extension Study to Assess the Long-Term Safety and Efficacy of CTP-543 in Adult Patients With Moderate to Severe Alopecia Areata
Brief Title: European Extension Study to Evaluate Safety and Efficacy of CTP-543 in Adults With Alopecia Areata
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Organization: Sun Pharmaceutical Industries Limited (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP543.5002; 2021-002365-18 (EudraCT Number)
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTP-543 (Experimental): Patients who previously completed a qualifying CTP-543 clinical trial
  Interventions: Drug: CTP-543

INTERVENTIONS:
Drug: CTP-543 — Twice daily dosing

SUMMARY:
The overall objectives of the study are to evaluate long-term safety of CTP-543 and to assess long-term effects of CTP-543 on treating hair loss in adult patients with chronic, severe alopecia areata. Patients from European sites who previously completed a qualifying CTP-543 clinical trial may participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Have completed 24 weeks of treatment in a previous qualifying CTP-543 clinical trial

Exclusion Criteria:

* Active scalp inflammation, psoriasis, or seborrheic dermatitis requiring topical treatment to the scalp, significant trauma to the scalp, or untreated actinic keratosis
* Females who are nursing, pregnant, or planning to become pregnant while in the study, and for 30 days after last dose of study medication
* Donation of blood at any point throughout the study and for 30 days after last dose of study medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- France (8):
  - Service de Dermatologie CHRU de Brest - Hopital Morvan, Brest, Finistere
  - Service de Dermatologie Centre Hospitalier Universitaire de Nice - Hopital Archet 2, Nice, Provence-Alpes-Côte d'Azur Region
  - CHU de Bordeaux, Hopital Saint-Andre, Bordeaux
  - Hopital Saint-Louis - GH De La Rochelle-Re-Aunis, La Rochelle
  - Hôpital La Timone-Dermatologie, Marseille
  - Hopital de l'Hotel Dieu - CHU de Nantes, Nantes
  - Hôpital Saint Louis, Centre de Santé Sabouraud, Paris
  - Centre Hospitalier Universitaire de Toulouse - Hopital Larrey, Toulouse
- Germany (7):
  - Universitätsklinikum Tübingen Universitäts-Hautklinik, Tübingen, Baden-Wüttermberg
  - Universitätsklinikum Erlangen, Hautklinik, Erlangen, Bavaria
  - Klinikum Rechts der Isar, Technische Universität München, Hautklinik, München, Bavaria
  - Klinik für Dermatologie, Venerologie und Allergologie, Frankfurt am Main, Hesse
  - Fachklinik Bad Bentheim, Bad Bentheim, Lower Saxony
  - Klinik für Dermatologie und Venerologie, Zentrale Studienkoordination für innovative Dermatologie (ZiD), Münster, North Rhine-Westphalia
  - Clinical Research Center for Hair and Skin Science, Dept of Dermatology, Charité Universitätsmedizin Berlin, Berlin
- Hungary (3):
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Bor-, Nemikortani es Onkodermatologiai Klinika, Pécs, Baranya
  - SZTE AOK Szent-Gyorgyi Albert Klinikai Kozpont, Borgyogyaszati es Allergologiai Klinika, Szeged, Csongrad-Csanad County
  - Semmelweis Egyetem AOK, Bor-, Nemikortani es Boronkologiai Klinika, Budapest, Pest County
- Poland (14):
  - Twoja Przychodnia Centrum Medyczne Nowa Sol, Nowa Sól, Lubusz Voivodeship
  - ETG Siedlce, Siedlce, Masovian Voivodeship
  - ETG Skierniewice, Skierniewice, Masovian Voivodeship
  - RCMed Oddzial w Sochaczewie, Sochaczew, Masovian Voivodeship
  - OT.CO Clinic Klinika Osipowicz & Turkowski sp. z o.o, Warsaw, Masovian Voivodeship
  - Carpe Diem Centrum Medycyny Estetycznej, Warsaw, Masovian Voivodeship
  - ETG Warszawa, Warsaw, Masovian Voivodeship
  - NZOZ Specjalistyczny Osrodek Dermatologiczny DERMAL, Bialystok
  - Vita Longa Sp.Zo.O, Katowice
  - Specjalistyczny Gabinet Dermatologiczny s.c., Krakow
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - My Clinic, Warsaw
  - Royalderm Agnieszka Nawrocka, Warsaw
  - WroMedica I. Bielicka, A. Strazalkowska s.c., Wroclaw
- Spain (7):
  - Hospital Clínic de Barcelona, Barcelona, Barcelona/Cataluña
  - Hospital del Mar, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid

RESULTS

PARTICIPANT FLOW:
Groups:
- CTP-543 8 mg BID: Participants received CTP-543 8 mg tablets, orally, twice a day
- CTP-543 12 mg BID: Participants received CTP-543 12 mg tablets, orally, twice a day
Period: Overall Study
Arm/Group | CTP-543 8 mg BID | CTP-543 12 mg BID
Started | 255 | 152
Completed | 201 | 127
Not Completed | 54 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CTP-543 8 mg BID | CTP-543 12 mg BID | Total
Number analyzed (Participants) | 255 | 152 | 407
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (12.41) | 38.2 (12.86) | 38.7 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181 | 89 | 270
  Male | 74 | 63 | 137
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 186 | 117 | 303
  Unknown or Not Reported | 62 | 30 | 92
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 193 | 121 | 314
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 62 | 30 | 92

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety
Time Frame: 108 weeks
Population: All subjects who received at least 1 dose of CTP-543 in this study. Subjects could be counted in both CTP-543 dose groups due to dose changes.
Measure: Count of Participants; unit: Participants
Arm/Group | CTP-543 8 mg BID | CTP-543 12 mg BID
Number analyzed (Participants) | 367 | 273
Participants | 308 | 224

2. Primary Outcome: Relative Change From Pre-zero Baseline in Total Severity of Alopecia Tool (SALT) Scores at Week 108
Description: SALT is a quantitative assessment of scalp hair loss with scores ranging from 0 (no scalp hair loss) to 100 (complete scalp hair loss). This outcome measures the relative Change from Pre-zero Baseline in Total SALT Scores. Relative change from baseline was defined as 100*(post-baseline value - baseline)/baseline.
Time Frame: 108 weeks
Population: Subjects received ≥1 dose of CTP-543 and ≥1 post-baseline SALT score. The 12 mg BID dose was removed per amended protocol; those on it were reduced to 8 mg BID and are shown in the (12→8 mg BID) group. Max 12 mg BID exposure was 81 weeks; by week 108, no subjects remained on it. Participant Flow reflects planned groups based on prior dose (active) or randomization (placebo). Analysis is based on initial treatment, then first new dose if changed.
Measure: Mean (Standard Deviation); unit: Percentage change
Groups:
- CTP-543 8 mg BID: Participants received CTP-543 8 mg tablets, orally, twice daily
- CTP-543 8 mg BID to CTP-543 12 mg BID: Participants received CTP-543 8 mg tablets orally twice daily as the first actual treatment, then 12 mg orally twice daily as the first dose change. After the 12 mg dose was removed from the study, participants either discontinued or reverted to 8 mg
- CTP-543 12 mg BID to CTP-543 8 mg BID: Participants received CTP-543 12 mg tablets orally, twice daily as the first actual treatment, then 8 mg orally, twice daily as the first dose change.
Arm/Group | CTP-543 8 mg BID | CTP-543 8 mg BID to CTP-543 12 mg BID | CTP-543 12 mg BID to CTP-543 8 mg BID
Number analyzed (Participants) | 97 | 48 | 99
Percentage change | -96.38 (8.790) | -88.57 (18.715) | -90.25 (18.860)

ADVERSE EVENTS:
Time Frame: 108 Weeks
Description: Subjects could be counted in both CTP-543 dose groups due to dose changes.
Arm/Group | CTP-543 8 mg BID | CTP-543 12 mg BID
All-Cause Mortality (participants affected / at risk) | 0/367 | 0/273
Serious Adverse Events (participants affected / at risk) | 16/367 | 5/273
Other Adverse Events (participants affected / at risk) | 176/367 | 127/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CTP-543 8 mg BID (N=367) | CTP-543 12 mg BID (N=273)
Bartholin's abscess (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis E (Infections and infestations) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (2) | 0 (0)
Gastric cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bartholin's cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intracranial hypotension (Nervous system disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CTP-543 8 mg BID (N=367) | CTP-543 12 mg BID (N=273)
Headache (Nervous system disorders) | 23 (27) | 9 (10)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 41 (46) | 29 (32)
Anaemia (Blood and lymphatic system disorders) | 13 (16) | 14 (17)
Thrombocytosis (Blood and lymphatic system disorders) | 20 (30) | 26 (28)
Weight increased (Investigations) | 14 (15) | 14 (14)
Nasopharyngitis (Infections and infestations) | 76 (118) | 48 (71)
Asymptomatic COVID-19 (Infections and infestations) | 83 (92) | 58 (65)
COVID-19 (Infections and infestations) | 78 (81) | 44 (46)
Upper respiratory tract infection (Infections and infestations) | 30 (50) | 14 (16)
Folliculitis (Infections and infestations) | 4 (4) | 14 (14)
Blood creatine phosphokinase increased (Investigations) | 42 (53) | 24 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-11-13): https://cdn.clinicaltrials.gov/large-docs/03/NCT05041803/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT05041803/SAP_001.pdf